CLINICAL TRIAL: NCT03578133
Title: A Cross-sectional Study Investigating the Causes of Pneumonia in Two Community Clinics in Two Yangon Townships, Myanmar
Brief Title: Causes of Pneumonia in Yangon
Status: Completed | Type: Observational
Sponsor: Myanmar Oxford Clinical Research Unit (Other)
Collaborators: Medical Action Myanmar (Other); Department of Medical Research, Myanmar (Unknown); Lao-Oxford-Mahosot Hospital Wellcome Trust Research Unit (Other)
Responsible Party: Sponsor
Other Study IDs: OXTREC 19-18
Record Dates: First submitted 2018-06-24; First posted 2018-07-05 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Melioidosis Pneumonia
Keywords: pneumonia; melioidosis; Myanmar; diagnosis
MeSH Terms: conditions — Pneumonia; Melioidosis; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: InBios® Active Melioidosis DetectTM-Lateral Flow Assay — Evaluation of a lateral flow assay for the detection of B.pseudomallei 6-deoxyheptan capsular polysaccharide antigen from sputum

SUMMARY:
This study will evaluate a new point of care diagnostic test for the diagnosis of melioidosis pneumonia in patients attending outpatient clinics in Yangon, Myanmar

DETAILED DESCRIPTION:
Melioidosis is caused by Burkholderia pseudomallei, a Gram-negative saprophytic environmental bacterium that is an important emerging tropical infection. There are an estimated 165,000 cases and 89,000 deaths world-wide each year. Eighty-four percent of cases are in SE Asia where mortality is 40%; far exceeding most recognised neglected tropical diseases. Pneumonia, secondary to either inhalation of B.pseudomallei or to bacteraemic spread to the lung is the commonest presentation (51%). Annually the highest burden (75%) of infection occurs in the rainy season in (75% in Thailand). Up to 80% patients have at least one recognised risk factor for melioidosis including; diabetes, alcohol-dependence, glucocorticoid therapy, chronic obstructive pulmonary disease (COPD), chronic renal disease and cancer. COPD and diabetes mellitus are amongst the top ten causes of death in Myanmar (2018). Patients with HIV have not been shown to have greater risk of B. pseudomallei than immunocompetent patients.

Melioidosis was discovered in Myanmar in 1911 by British pathologist Alfred Whitmore and his assistant CS Krishnaswami. Yet since 1949 there have been few published cases. Under-reporting is partly due to difficulty in diagnosing melioidosis. Clinical and radiological findings are indistinguishable from tuberculosis. Laboratory diagnosis is challenging, lack of facilities, expertise and awareness of B.pseudomallei results in missed diagnostic opportunities.

Culture is the gold-standard diagnostic method but requires appropriate facilities and expertise which are not readily available in many developing countries like Myanmar. A rapid diagnostic (RDT) test has been developed for low resource settings that has been evaluated in Laos and India. The InBios® Active Melioidosis DetectTM-Lateral Flow Assay (AMD-LFA) detects B.pseudomallei 6-deoxyheptan capsular polysaccharide antigen. Shaw et al demonstrated sensitivity 85.71% (CI:74.61% to 93.25%) and specificity 93.62% (CI:88.23% to 97.04%), with positive predictive value of 85.71% (CI: 75.98% to 91.92%) compared to culture. We propose to evaluate this test for the diagnosis of melioidosis pneumonia in Myanmar.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. Reported fever or axillary temperature > 37.5 °C
3. Productive cough
4. Written informed consent

Exclusion Criteria:

1. Inability to provide a sputum specimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population investigated will be patients attending two non-governmental organisation community clinics in the most deprived areas of Yangon, Myanmar
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a positive B.pseudomallei culture result | January 2019
  Number of patients with a positive sputum culture for B.pseudomallei expressed as a proportion of all patients
1) Sensitivity, specificity, positive predictive value, negative predictive value of the RDT compared to culture | January 2019
  Using culture as the gold-standard the performance of the lateral flow assay will be assessed

SECONDARY OUTCOMES:
Proportion of patients diagnosed with tuberculosis (TB) including multidrug resistant TB | January 2019
  Proportion of enrolled participants with a positive GeneXpert MTB/RIF test on sputum
Proportion of patients diagnosed with Influenza A/B | March 2019
  Proportion of enrolled participants with a positive Xpert Flu test on nasopharyngeal swab

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Ashley, Dr, Principal Investigator — Myanmar Oxford Clinical Research Unit; Frank Smithuis, Prof, Principal Investigator — Myanmar Oxford Clinical Research Unit and Medical Action Myanmar; Clare Warrell, Dr, Study Director — Myanmar Oxford Clinical Research Unit and Medical Action Myanmar; David Dance, Prof, Study Director — Lao-Oxford-Mahosot Hospital Wellcome Trust Research Unit; Ni Ni Tun, Dr, Study Director — Medical Action Myanmar; Mo Mo Win, Dr, Study Director — Department of Medical Research, Myanmar; Alistair McLean, Dr, Study Director — Myanmar Oxford Clinical Research Unit; Kyaw Soe, Study Director — Myanmar Oxford Clinical Research Unit
Locations (1):
- Medical Action Myanmar Clinics, Yangon, Burma

REFERENCES:
- [Background] Limmathurotsakul D, Golding N, Dance DA, Messina JP, Pigott DM, Moyes CL, Rolim DB, Bertherat E, Day NP, Peacock SJ, Hay SI. Predicted global distribution of Burkholderia pseudomallei and burden of melioidosis. Nat Microbiol. 2016 Jan 11;1:15008. doi: 10.1038/nmicrobiol.2015.8. PMID 27571754
- [Background] Houghton RL, Reed DE, Hubbard MA, Dillon MJ, Chen H, Currie BJ, Mayo M, Sarovich DS, Theobald V, Limmathurotsakul D, Wongsuvan G, Chantratita N, Peacock SJ, Hoffmaster AR, Duval B, Brett PJ, Burtnick MN, Aucoin DP. Development of a prototype lateral flow immunoassay (LFI) for the rapid diagnosis of melioidosis. PLoS Negl Trop Dis. 2014 Mar 20;8(3):e2727. doi: 10.1371/journal.pntd.0002727. eCollection 2014 Mar. PMID 24651568
- [Background] Chierakul W, Wuthiekanun V, Chaowagul W, Amornchai P, Cheng AC, White NJ, Day NP, Peacock SJ. Short report: disease severity and outcome of melioidosis in HIV coinfected individuals. Am J Trop Med Hyg. 2005 Dec;73(6):1165-6. PMID 16354832
- [Background] Shaw T, Tellapragada C, Ke V, AuCoin DP, Mukhopadhyay C. Performance evaluation of Active Melioidosis Detect-Lateral Flow Assay (AMD-LFA) for diagnosis of melioidosis in endemic settings with limited resources. PLoS One. 2018 Mar 26;13(3):e0194595. doi: 10.1371/journal.pone.0194595. eCollection 2018. PMID 29579128
- [Background] Woods KL, Boutthasavong L, NicFhogartaigh C, Lee SJ, Davong V, AuCoin DP, Dance DAB. Evaluation of a Rapid Diagnostic Test for Detection of Burkholderia pseudomallei in the Lao People's Democratic Republic. J Clin Microbiol. 2018 Jun 25;56(7):e02002-17. doi: 10.1128/JCM.02002-17. Print 2018 Jul. PMID 29720430
- [Background] Wiersinga WJ, Currie BJ, Peacock SJ. Melioidosis. N Engl J Med. 2012 Sep 13;367(11):1035-44. doi: 10.1056/NEJMra1204699. No abstract available. PMID 22970946